CLINICAL TRIAL: NCT05592639
Title: Videoendoscopic Radical Inguinal Lymphadenectomy Versus Open Radical Inguinal Lymphadenectomy in Patients With Penile Cancer: a Feasibility Randomised Controlled Trial
Brief Title: VideoEndoscopic Radical Inguinal Lymphadenectomy for Penile Cancer
Acronym: VELRAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: The Christie NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 130062
Record Dates: First submitted 2022-10-13; First posted 2022-10-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Penile Cancer; Inguinal Lymphadenopathy; Melanoma
MeSH Terms: conditions — Penile Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videoendoscopic Inguinal Lymphadenectomy (Active Comparator): Removal of inguinal nodes using Videoendoscopic Inguinal Lymphadenectomy
  Interventions: Procedure: Videoendoscopic radical inguinal lymphadenectomy or open radical inguinal lymphadenectomy
- Open Inguinal Lymphadenectomy (Other): Removal of inguinal nodes using Open radical inguinal lymphadenectomy
  Interventions: Procedure: Videoendoscopic radical inguinal lymphadenectomy or open radical inguinal lymphadenectomy

INTERVENTIONS:
Procedure: Videoendoscopic radical inguinal lymphadenectomy or open radical inguinal lymphadenectomy — Intervention is a Videoendoscopic radical inguinal lymphadenectomy (VEIL) which is a surgical technique utilised in removing inguinal lymph nodes.

SUMMARY:
Assess the feasibility of performing a RCT comparing videoendoscopic radical inguinal lymphadenectomy versus open radical inguinal lymphadenectomy in men diagnosed with genital cancer requiring inguinal lymphadenectomy, and determine the design of such an RCT.

DETAILED DESCRIPTION:
There is increasing interest in using videoendoscopic inguinal lymph node dissection (ILND) as an alternative to open ILND. Videoendoscopic inguinal lymphadenectomy (VEIL) may decrease complications compared to open ILND and provide equivalent short-term oncological outcomes.

As yet, there have been no randomised-controlled trials (RCTs) comparing these procedures.

VELRAD aims to assess the feasibility of performing a RCT comparing VEIL and open ILND. This will be measured by recruitment rate, the acceptability of the trial design and intervention to clinical stage and patients. Investigators will also collect qualitative data on why patients did or did not agree to be randomised

ELIGIBILITY:
Inclusion Criteria:

1. People requiring inguinal lymphadenectomy i.e.

   1. Patients with squamous cell carcinoma or mucosal melanoma of the penis > T1bG2 or patients with male genital cancer requiring inguinal lymphadenectomy
   2. Patients unsuitable for dynamic sentinel node biopsy (DSNB) with impalpable nodes: previous penectomy or non-visualisation at previous DSNB
   3. Previous DSNB with metastatic inguinal nodes on histology or FNA positive nodes on cytology who require a completion radical inguinal lymphadenectomy
   4. Small volume palpable inguinal lymph nodes (< 2 cm on CT) not fixed to skin
2. Age > 18 years

Exclusion Criteria:

1. Unfit for surgery
2. People unlikely to benefit from lymphadenectomy because of advanced cancer
3. Those with palpable inguinal lymph nodes fixed to skin or adjacent structures
4. Does not want to participate in the trial or unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Ability to recruit patients | 18 months
  Ability to recruit patients at the selected sites (recruitment rate)

CONTACTS AND LOCATIONS:
Overall Officials: Asif Muneer, MD, Principal Investigator — University College, London
Locations (1):
- University College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang S, Akers C, Alnajjar H, Ayres B, Baldini C, Embleton-Thirsk A, Gurusamy K, Hadway P, Kumar V, Lau M, Nigam R, Pang K, Parnham A, Pizzo E, Ranieri V, Rees R, Sangar V, Wadke A, Williams N, Muneer A. A study protocol for a feasibility randomised controlled trial investigating videoendoscopic radical inguinal lymphadenectomy versus open radical inguinal lymphadenectomy in patients with penile cancer (VELRAD). Pilot Feasibility Stud. 2024 Apr 10;10(1):61. doi: 10.1186/s40814-024-01474-8. PMID 38600541